CLINICAL TRIAL: NCT04990869
Title: Effects of Nicotinamide Riboside on the Airway Inflammation of Older Adults With COPD: A Randomized, Double-blind, Placebo-controlled Clinical Trial (NR-COPD)
Brief Title: Inflammation in COPD and the Effect of Nicotinamide Riboside
Acronym: ICON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Bispebjerg Hospital (Other); Elysium Health (Industry)
Responsible Party: Principal Investigator, Morten Scheibye-Knudsen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NR-COPD
Record Dates: First submitted 2021-06-28; First posted 2021-08-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COPD-NR (Experimental): COPD patients receiving Nicotinamide Riboside
  Interventions: Dietary Supplement: Nicotinamide Riboside
- COPD-placebo (Placebo Comparator): COPD patients receiving placebo
  Interventions: Dietary Supplement: Placebo
- Control-NR (Experimental): Lung-healthy controls receiving Nicotinamide Riboside
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Control-placebo (Placebo Comparator): Lung-healthy controls receiving placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — The patients will receive 1 g of Nicotinamide Riboside or placebo orally every morning and evening for 6 weeks.
  Arms: COPD-NR; Control-NR
Dietary Supplement: Placebo — Placebo
  Arms: COPD-placebo; Control-placebo

SUMMARY:
The aim of this study is to investigate if nicotinamide riboside can reduce the airways inflammation associated with chronic obstructive pulmonary disease (COPD) in patients aged 60 or older. A major event in aging is the loss of the central metabolite nicotinamide adenine dinucleotide (NAD+) that appear to be important in the proinflammatory environment that occur during aging. Notably, recent work suggest that aging can be ameliorated by even a short-term treatment of the NAD+ precursor nicotinamide riboside. Nicotinamide riboside has recently been shown to be able to return aging tissues to a younger state even after short term treatment. This vitamin B3- analog is naturally occurring, is readily taken up through oral administration and has been tested in human trials with few side effects. The investigators hypothesize that six weeks of nicotinamide riboside supplementation reduces interleukin-8 measured in sputum from COPD patients. Further, it is hypothesized that augmentation of NAD+ in COPD patients might alleviate symptoms through activation of sirtuins.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major problem that affect more and more people worldwide with over three million deaths reported every year. COPD has been described as a disease of accelerated lung aging and is associated with oxidative stress and an increased inflammatory response to for instance viral infections. Therefore, in the current pandemic COPD patients are considered at high risk of COVID-19-related death and interventions in this group are crucial.

A major event in aging is the loss of nicotinamide adenine dinucleotide (NAD+)-a loss which may be important in promoting the pro-inflammatory environment that occur with aging and therefore possibly COPD. Indeed, NAD+ is emerging as a central metabolic molecule involved in multiple age-related pathways including inflammation and metabolic control. Recently, it was shown that age-associated NAD+ loss is due to macrophage M1-polarization, suggesting that NAD+ is required for macrophage activation, an event that is involved in the pulmonary inflammatory response. In humans, the therapeutic potential of boosting NAD+ levels through supplementation with one of its more bioavailable precursors has therefore gained attention.

Nicotinamide riboside (NR) is a NAD+ precursor and recent work suggests that aging can be ameliorated by even short-term treatment with NR. This vitamin B3-analog is naturally occurring, is readily taken up through oral administration and has been tested in human trials with few side effects. Notably, NR treatment in humans decreases circulating markers of inflammation. In addition, NAD+ replenishment may facilitate overall greater resilience of older patients considering the anti-aging effects of NR allowing these patients to better cope with infections. Interestingly, NR has been shown to return aging tissues to a younger state, possibly through augmentation of the sirtuin enzyme family-known to play an important role in almost all cellular functions. COPD patients have reduced sirtuin levels in the airways likely due to oxidative stress. Because sirtuins are NAD+-dependent, supplementation with NR could serve as a treatment option for patients with COPD through activation of sirtuins. In addition, NAD+ replenishment may facilitate overall greater resilience of older patients considering the anti-aging effects of nicotinamide riboside allowing these patients to better cope with infections.

The chosen dosage is 2 g per day given orally. This dose has been shown to be safe and tolerated. The dose will be split in two with ingestion of 1 g in the morning and 1 g in the evening. NR is a naturally occurring vitamin B3 analog produced by yeast and found in multiple food products at low concentration. Many organisms including humans cannot produce NR but have instead evolved methods to convert this into the central redox modulator NAD+.

The efficacy and safety of NR supplementation has been tested in a number of studies in both healthy middle-aged and older adults and in patients suffering from metabolic disease. Since this is a natural compound widely found in nature no subjects have yet developed allergic responses to the molecule, and repeated doses of up to 2 g orally per day have demonstrated an acceptable safety profile. No treatment-emergent adverse events have so far been reported for NR.

Older adults (age ≥ 60 years) with a diagnosis of COPD will be recruited from the Respiratory Medicine and Emergency departments at Bispebjerg Hospital, Denmark, and through advertisements on online websites (e.g. www.lungeforskning.dk). Lung-healthy controls will be recruited through online websites (e.g. www.forsøgsperson.dk). Potential participants will be asked if they want to participate in this trial and informed about the study procedures. If they agree and if they meet the inclusion and not the exclusion criteria, the subjects will be randomized to either the NR or placebo group. All subjects that give informed consent to participate will receive a study identification number.

Study endpoints will be assessed at baseline, after the 6-week treatment and follow-up after 18 weeks. Telephone follow-up will be conducted after 58 weeks. Endpoints include airway inflammation measured in sputum, untargeted RNA sequencing of nasal epithelial cells, DNA methylation and untargeted metabolomics in peripheral mononucleated cells, circulating inflammatory markers and NAD+ levels in whole-blood, in addition to clinical outcomes such as lung function (spirometry), chest x-ray and questionnaires.

ELIGIBILITY:
Inclusion Criteria COPD patients:

1. Written informed consent.
2. Age 60 or older.
3. A body mass index (BMI) between 18.5-40.0 kg·m-2 and a weight ≥ 40 kg at enrolment.
4. A diagnosis of chronic obstructive pulmonary disease (FEV1/FVC < 0.7).
5. Smoking history of at least 10 pack years, but currently ex-smoker.
6. Not using any inhalation steroids.
7. A worsening of symptoms in relation to respiratory infections.
8. Eosinophil count < 0.3 at inclusion or within 3 months.

Exclusion Criteria COPD patients:

1. Exacerbation of COPD or severe airway infection within the last two months.
2. Chronic use of supplements containing vitamin B or NR.
3. Planned surgery during the course of the trial.
4. Dementia/cognitive impairment or symptomatic psychiatric illness.
5. Cancer diagnosis within last 5 years.
6. Inability to speak and read Danish.
7. Unwillingness or inability to follow the procedures outlined in the protocol.
8. Concurrent enrollment in another clinical study involving an investigational treatment.

Inclusion Criteria Controls:

1. Written informed consent.
2. Age-, sex- and BMI-matched with COPD patients.
3. No history of lung disease.
4. Never-smoker.

Exclusion Criteria Controls:

1. Chronic use of supplements containing vitamin B or NR.
2. Planned surgery during the course of the trial.
3. Dementia/cognitive impairment or symptomatic psychiatric illness.
4. Cancer diagnosis within last 5 years.
5. Inability to speak and read Danish.
6. Unwillingness or inability to follow the procedures outlined in the protocol.
7. Concurrent enrollment in another clinical study involving an investigational treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Interleukin-8 | 6 weeks
  Measured in sputum

SECONDARY OUTCOMES:
NAD+ levels | 6 weeks
  Measured in whole-blood
Interleukin-6 | 6 weeks
  Measured in plasma
Interleukin-10 | 6 weeks
  Measured in plasma
Tumor necrosis factor alpha | 6 weeks
  Measured in plasma
C-reactive protein | 6 weeks
  Measured in plasma
Matrix metalloproteinase-9 | 6 weeks
  Measured in plasma

OTHER OUTCOMES:
Untargeted metabolomics | 6 weeks
  Measured in peripheral blood mononucleated cells
Untargeted RNA sequencing | 6 weeks
  Measured in nasal epithelial cells
DNA methylation | 6 weeks
  Measured in peripheral blood mononucleated cells

CONTACTS AND LOCATIONS:
Overall Officials: Morten Scheibye-Knudsen, MD/DMSc(PhD), Principal Investigator — University of Copenhagen
Locations (1):
- Respiratory Research Unit, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Norheim KL, Ben Ezra M, Heckenbach I, Andreasson LM, Eriksen LL, Dyhre-Petersen N, Damgaard MV, Berglind M, Pricolo L, Sampson D, Dellinger RW, Sverrild A, Treebak JT, Ditlev SB, Porsbjerg C, Scheibye-Knudsen M. Effect of nicotinamide riboside on airway inflammation in COPD: a randomized, placebo-controlled trial. Nat Aging. 2024 Dec;4(12):1772-1781. doi: 10.1038/s43587-024-00758-1. Epub 2024 Nov 15. PMID 39548320